CLINICAL TRIAL: NCT02222688
Title: A Phase I Clinical Trial to Determine the Safety and Tolerability of UC-961 (Cirmtuzumab), an Anti-ROR1 Monoclonal Antibody, for the Treatment of Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia Who Are Ineligible for Chemotherapy
Brief Title: UC-961 (Cirmtuzumab) in Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Thomas Kipps (Other)
Responsible Party: Sponsor-Investigator, Thomas Kipps, Deputy Director of Research Operations, Moores Cancer Center, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: #140141
Record Dates: First submitted 2014-08-19; First posted 2014-08-21 (Estimated); Results first posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: cancer; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — cirmtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cirmtuzumab 0.015 - 0.03 mg/kg (Experimental): Cohort 1: Cirmtuzumab 0.015 mg/kg for two 14-day cycles followed by cirmtuzumab 0.03 mg/kg for two 14-day cycles via intravenous (IV) infusion
  Interventions: Drug: cirmtuzumab
- Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg (Experimental): Cohort 2: Cirmtuzumab 0.06 mg/kg for one 14-day cycle, followed by cirmtuzumab 0.12 mg/kg for one 14-day cycle, followed by 0.24 mg/kg for two 14-day cycles via IV infusion
  Interventions: Drug: cirmtuzumab
- Cirmtuzumab 0.5 - 1.0 mg/kg (Experimental): Cohort 3: Cirmtuzumab 0.5 mg/kg for one 14-day cycle, followed by cirmtuzumab 1.0 mg/kg for three 14-day cycles via IV infusion
  Interventions: Drug: cirmtuzumab
- Cirmtuzumab 2.0 - 4.0 mg/kg (Experimental): Cohort 4: Cirmtuzumab 2.0 mg/kg for two 14-day cycles, followed by cirmtuzumab 4.0 mg/kg for two 14-day cycles via IV infusion
  Interventions: Drug: cirmtuzumab
- Cirmtuzumab 8 mg/kg (Experimental): Cohort 5: Cirmtuzumab 8 mg/kg for four 14-day cycles via IV infusion
  Interventions: Drug: cirmtuzumab
- Cirmtuzumab 16 mg/kg (Experimental): Cohort 6: Cirmtuzumab 16 mg/kg for four 14-day cycles (or maximum 2000 mg) via IV infusion
  Interventions: Drug: cirmtuzumab
- Cirmtuzumab 20 mg/kg (Experimental): Cohort 7: Cirmtuzumab 20 mg/kg for four 14-day cycles (or maximum 2000 mg)
  Interventions: Drug: cirmtuzumab

INTERVENTIONS:
Drug: cirmtuzumab
  Other Names: UC-961

SUMMARY:
The purpose of the study is to investigate the safety of the investigational agent, cirmtuzumab. Cirmtuzumab is a monoclonal antibody drug designed to attach to a protein, called ROR1, on the surface of chronic lymphocytic leukemia (CLL) cells to block cell growth and survival. ROR1 is rarely expressed on healthy cells so the idea is to preferentially get rid of the cancer cells. Although there is evidence in laboratory animals that cirmtuzumab can decrease the number of CLL cells, the investigators do not know if this will work in humans. This drug will be given to humans for the first time in this study. Therefore, the goal of this study is to see if cirmtuzumab is safe and tolerated in study participants.

DETAILED DESCRIPTION:
This is a first in human, open-label single institution, Phase I dose escalation study of in patients with relapsed or refractory CLL. Treatment cycle (14 days) will consist of cirmtuzumab administered intravenously on a bi-weekly (every two weeks) schedule for a total of 4 doses. Eight dose cohorts (of 3 to 6 patients in size) plus an expansion cohort of 6 patients are planned. In the first 4 dose cohorts, there is intra-patient dose escalation to monitor for acute toxicities, such as tumor lysis syndrome.

A cycle may be repeated every 14 days if the patient has at least stable disease by clinical examination (or interim response assessment) and has again met hematologic, renal, and hepatic laboratory parameters as defined in the eligibility section, and is without ongoing Grade 3 non-hematologic or Grade 4 hematologic toxicities attributable to cirmtuzumab. The total duration of study drug administration is 4 cycles. Each cycle consists of clinical and laboratory evaluation on Day 1 and safety assessments on Days 3 and 8.

ELIGIBILITY:
INCLUSION CRITERIA:

* Clinical and phenotypic verification of B cell CLL and measurable disease. Immunophenotyping of the leukemic cells must demonstrate a monoclonal B cell population with immunophenotype consistent with CLL.
* Relapsed or refractory disease, defined by failure to achieve a partial response within 6 months of initiation of therapy, or a 50% increase of baseline disease measurements after achieving a clinical response.
* Not amenable to approved therapies.
* Prior Therapy: Must have progressed after purine-analog or alkylator based therapy, or be considered inappropriate for chemo-immunotherapy due to one of the following:

  * Del 17p, which is associated with poor response to chemo-immunotherapy, or
  * Age greater than 70, or
  * Age greater than 65 with one of the following:
  * Grade ≥ 3 neutropenia, anemia, or thrombocytopenia attributable to cumulative myelotoxicity from prior administration of cytotoxic agents (as documented by bone marrow biopsy obtained since last prior therapy), or
  * Clinically apparent autoimmune cytopenia which may be exacerbated by fludarabine therapy, or
  * Estimated creatinine clearance (eCCr) <70 mL/min (as determined by the Cockcroft-Gault method), or
  * Eastern Cooperative Oncology Group (ECOG) performance status greater than 0.
* Has recovered from the toxic effects of prior therapy to their clinical baseline.
* Women of childbearing potential must agree not to become pregnant for the duration of the study. Both men and women must agree to use a barrier method of contraception for the duration of the study and until 10 weeks after the final dose of cirmtuzumab.
* Subjects must have at least one of the following indications for treatment:

  * Symptomatic or progressive splenomegaly;
  * Symptomatic lymph nodes, nodal clusters, or progressive lymphadenopathy;
  * Progressive anemia (hemoglobin ≤ 11 g/dL);
  * Progressive thrombocytopenia (platelets ≤ 100 x 10^9/L);
  * Weight loss > 10% body weight over the preceding 6 month period;
  * Fatigue attributable to CLL;
  * Fever or night sweats for > 2 weeks without evidence of infection;
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period or an anticipated doubling time of less than 12 months.
* Subjects must have an ECOG performance status of 0-2.
* Adequate hematologic function
* Adequate renal function
* Adequate hepatic function
* Adequate coagulation tests

EXCLUSION CRITERIA:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies.
* Patients who are currently receiving another investigational agent are excluded.
* Patients who have had chemotherapy (e.g., purine analogues, alkylating agents), immunotherapy, radiation therapy, or participation in any investigational drug treatment within 4 weeks of initiation of UC-961 or at any time during the study.
* Patients who have had prior (within 8 weeks of initiation of UC-961) or concurrent antibody therapy directed against CLL (i.e., Rituxan® and Campath®).
* Current infection requiring parenteral antibiotics.
* Active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV).
* Concurrent malignancy or prior malignancy within the previous 3 years (other than completely resected carcinoma in situ, prostate cancer, or localized non-melanoma skin cancer).
* Known central nervous system (CNS) involvement by malignancy.
* Untreated autoimmunity such as autoimmune hemolytic anemia, or immune thrombocytopenia.
* Uncompensated hypothyroidism (defined as thyroid-stimulating hormone (TSH) greater than 2x upper limit of normal not treated with replacement hormone).
* Presence of more than 55% pro-lymphocytes in peripheral blood. Patients with Richter's transformation are not excluded.
* Insufficient recovery from surgical-related trauma or wound healing.
* Impaired cardiac function including any of the following:

  * Myocardial infarction within 6 months of starting study drug;
  * A past medical history of clinically significant ECG abnormalities, including QTc 481 milliseconds or greater;
  * Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08-08 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona Jamieson, M.D., Ph.D., Principal Investigator — University of California Medical Center; Michael Choi, M.D., Principal Investigator — University of Calilfornia Medical Center
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

REFERENCES:
- [Result] Choi MY, Widhopf GF 2nd, Ghia EM, Kidwell RL, Hasan MK, Yu J, Rassenti LZ, Chen L, Chen Y, Pittman E, Pu M, Messer K, Prussak CE, Castro JE, Jamieson C, Kipps TJ. Phase I Trial: Cirmtuzumab Inhibits ROR1 Signaling and Stemness Signatures in Patients with Chronic Lymphocytic Leukemia. Cell Stem Cell. 2018 Jun 1;22(6):951-959.e3. doi: 10.1016/j.stem.2018.05.018. PMID 29859176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled into the study between August 2014 and September 2017 and included patients seen in the UCSD Health system.
Pre-assignment Details: Twenty-seven subjects were treated with cirmtuzumab and are included in the primary outcome analysis. One subject was enrolled into the trial twice; first in Cohort 1 and then again in Cohort 4 and is counted once for reporting of the baseline characteristics.
Groups:
- Cimrtuzumab 2.0 - 4.0 mg/kg: Cohort 4: Cirmtuzumab 2.0 mg/kg for two 14-day cycles, followed by cirmtuzumab 4.0 mg/kg for two 14-day cycles via IV infusion
Period: Overall Study
Arm/Group | Cirmtuzumab 0.015 - 0.03 mg/kg | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg | Cirmtuzumab 0.5 - 1.0 mg/kg | Cimrtuzumab 2.0 - 4.0 mg/kg | Cirmtuzumab 8 mg/kg | Cirmtuzumab 16 mg/kg | Cirmtuzumab 20 mg/kg
Started | 4 | 3 | 3 | 5 | 3 | 3 | 6
Completed | 3 | 3 | 3 | 3 | 2 | 3 | 5
Not Completed | 1 | 0 | 0 | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 1 | 0 | 1
Not completed — Disease progression | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Twenty-seven subjects were treated with cirmtuzumab and are included in the primary outcome analysis. One subject was enrolled into the trial twice; first in Cohort 1 and then again in Cohort 4 and is counted twice for the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cirmtuzumab 0.015 - 0.03 mg/kg | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg | Cirmtuzumab 0.5 - 1.0 mg/kg | Cirmtuzumab 2.0 - 4.0 mg/kg | Cirmtuzumab 8 mg/kg | Cirmtuzumab 16 mg/kg | Cirmtuzumab 20 mg/kg | Total
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 3 | 6 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 5
  >=65 years | 4 | 2 | 2 | 4 | 3 | 2 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.75 (1.5) | 70.67 (11.68) | 66.67 (3.51) | 69.4 (7.23) | 70 (2.65) | 71.67 (9.29) | 77.33 (8.78) | 71.81 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 3 | 1 | 1 | 4 | 13
  Male | 2 | 1 | 3 | 2 | 2 | 2 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 3 | 5 | 3 | 3 | 6 | 27
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 2 | 5 | 3 | 2 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 5 | 3 | 3 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) or Biologically Active Dose of Cirmtuzumab
Description: The MTD is defined as the highest dose studied at which no more than one in six patients experience a dose-limiting toxicity (DLT) during the DLT observation period. The biologically active dose will be determined at a dose below or equal to the MTD upon review of the the study data; the final determination will also consider any cumulative or delayed toxicity.
Time Frame: 1 year
Measure: Number; unit: mg/kg
Groups:
- All Participants: All participants who received any treatment with cirmtuzumab
Arm/Group | All Participants
Number analyzed (Participants) | 27
mg/kg | 20

2. Primary Outcome: Rate of Dose Limiting Toxicities (DLTs)
Description: The occurrence of any of the following adverse events considered to be possibly, probably, or definitely related to cirmtuzumab within the DLT observation period (56 days from the first infusion for cohorts with intrapatient dose escalation, and 28 days of the start investigational treatment for cohorts without intrapatient dose escalation):
  1. Grade 3 or greater non-hematologic toxicity with the exception of Grade 3 infusion reaction.
  2. Grade 4 neutropenia lasting more than 5 days despite appropriate medical management.
  3. Grade 4 thrombocytopenia or grade 3 thrombocytopenia with bleeding or any requirement for platelets transfusion.
  4. Grade 3 or greater febrile neutropenia (temperature ≥ 38.5ºC).
  5. Grade 4 anemia unexplained by underlying disease.
  6. Any AE requiring a dose delay of greater than 14 days.
  7. Patients with baseline cytopenias or starting blood counts in the grade 2 range are evaluable for hematologic DLT.
Time Frame: The DLT observation period is 56 days from the start of the first infusion for the intra-patient dosing cohorts and 28 days after the start of the first infusion for subsequent dosing cohorts
Measure: Number; unit: Occurrence of DLTs
Arm/Group | Cirmtuzumab 0.015 - 0.03 mg/kg | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg | Cirmtuzumab 0.5 - 1.0 mg/kg | Cirmtuzumab 2.0 - 4.0 mg/kg | Cirmtuzumab 8 mg/kg | Cirmtuzumab 16 mg/kg | Cirmtuzumab 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 3 | 6
Occurrence of DLTs | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Safety and Tolerability of UC-961 by Ongoing Evaluation of AEs.
Description: Treatment emergent adverse events (description, timing, CTCAE grade, severity, seriousness, and relatedness)
Time Frame: From the start of investigational treatment to completion of follow-up, an average of 33 weeks
Measure: Number; unit: Treatment emergent AEs
Arm/Group | Cirmtuzumab 0.015 - 0.03 mg/kg | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg | Cirmtuzumab 0.5 - 1.0 mg/kg | Cirmtuzumab 2.0 - 4.0 mg/kg | Cirmtuzumab 8 mg/kg | Cirmtuzumab 16 mg/kg | Cirmtuzumab 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 3 | 6
Treatment emergent AEs | 20 | 37 | 15 | 31 | 17 | 34 | 46

4. Secondary Outcome: Clinical Activity Determined by the International Working Group in CLL (iwCLL) Criteria
Description: Clinical response [stable disease (SD) or progressive disease (PD)] defined by iwCLL criteria including clinical, hematological, and bone marrow features for a period of at least 2 months from completion of therapy
Time Frame: From baseline visit to response assessment visit at 56 days after final cirmtuzumab infusion, an average of 52 days
Population: Evaluable subjects or those who completed 4 cycles of cirmtuzumab
Measure: Number; unit: participants
Arm/Group | Cirmtuzumab 0.015 - 0.03 mg/kg | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg | Cirmtuzumab 0.5 - 1.0 mg/kg | Cirmtuzumab 2.0 - 4.0 mg/kg | Cirmtuzumab 8 mg/kg | Cirmtuzumab 16 mg/kg | Cirmtuzumab 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2 | 3 | 5
participants
  Stable Disease | 0 | 0 | 1 | 0 | 1 | 1 | 2
  Progressive Disease | 3 | 3 | 2 | 3 | 1 | 2 | 3

5. Secondary Outcome: Progression Free Survival as Determined by iwCLL Criteria
Description: The duration of time from the start of study treatment until objective tumor progression or death
Time Frame: From start of treatment until objective tumor progression or death
Measure: Mean (Full Range); unit: Weeks
Groups:
- Cirmtuzumab 20 mg/kg: Cohort 7: Cirmtuzumab 20 mg/kg for four 14-day cycles (or maximum 2000 mg) via IV infusion
Arm/Group | Cirmtuzumab 0.015 - 0.03 mg/kg | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg | Cirmtuzumab 0.5 - 1.0 mg/kg | Cirmtuzumab 2.0 - 4.0 mg/kg | Cirmtuzumab 8 mg/kg | Cirmtuzumab 16 mg/kg | Cirmtuzumab 20 mg/kg
Number analyzed (Participants) | 4 | 3 | 3 | 5 | 3 | 3 | 6
Weeks | 29.5 [2.0 to 79.9] | 27.6 [10.5 to 54.2] | 24.5 [18.5 to 32] | 36.6 [1 to 136] | 25.4 [4 to 42.2] | 26.2 [20.5 to 29] | 19.9 [5.2 to 56.3]

ADVERSE EVENTS:
Time Frame: Adverse events collected from the start of the first infusion of cirmtuzumab to the last subject's final visit in long-term follow-up (on average 3 years 8 months)
Description: Note that some patients elected to enroll in extension study (ClinicalTrails.gov record #NCT02860676) and therefor the cut-off date for some may be the date patient was first treated on extension protocol. Timeframe for this result therefore difficult to reconcile as asked to report here.
  Note no deaths observed during the timeframe of the study observation period.
Arm/Group | Cirmtuzumab 0.015 - 0.03 mg/kg | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg | Cirmtuzumab 0.5 - 1.0 mg/kg | Cimrtuzumab 2.0 - 4.0 mg/kg | Cirmtuzumab 8 mg/kg | Cirmtuzumab 16 mg/kg | Cirmtuzumab 20 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/5 | 0/3 | 0/3 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/3 | 0/5 | 0/3 | 1/3 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 5/5 | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cirmtuzumab 0.015 - 0.03 mg/kg (N=4) | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg (N=3) | Cirmtuzumab 0.5 - 1.0 mg/kg (N=3) | Cimrtuzumab 2.0 - 4.0 mg/kg (N=5) | Cirmtuzumab 8 mg/kg (N=3) | Cirmtuzumab 16 mg/kg (N=3) | Cirmtuzumab 20 mg/kg (N=6)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Grade 3, assessed as unlikely related to investigational drug
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 2, assessed as not related to investigational drug
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Grade 3, assessed as unlikely related to investigational drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cirmtuzumab 0.015 - 0.03 mg/kg (N=4) | Cirmtuzumab 0.06 - 0.12 - 0.24 mg/kg (N=3) | Cirmtuzumab 0.5 - 1.0 mg/kg (N=3) | Cimrtuzumab 2.0 - 4.0 mg/kg (N=5) | Cirmtuzumab 8 mg/kg (N=3) | Cirmtuzumab 16 mg/kg (N=3) | Cirmtuzumab 20 mg/kg (N=6)
Anemia (Blood and lymphatic system disorders) | 4 (6) | 3 (12) | 3 (9) | 3 (9) | 3 (10) | 3 (14) | 4 (10)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eye disorders - other (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Floater (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal disorders - other (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Flu-like symptoms (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 3 (6) | 1 (1)
Serum amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 4 (13) | 2 (9) | 2 (4) | 4 (8) | 3 (5) | 2 (7) | 1 (11)
Neutropenia (Investigations) | 1 (4) | 2 (7) | 2 (4) | 2 (2) | 2 (3) | 2 (10) | 1 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3)
Parasthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Some patients enrolled in extension study (#NCT02860676)& cut-off date for AE observation may be date patient was first treated on extension, therefor AE Timeframe period difficult to reconcile. 0 deaths observed during study observation period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT02222688/Prot_SAP_000.pdf